CLINICAL TRIAL: NCT02722408
Title: A Phase 2 Open-Label, Dose-Finding Study to Assess the Efficacy, Safety, and Tolerability of Gemcabene in Patients With Homozygous Familial Hypercholesterolemia on Stable, Lipid Lowering Therapy (COBALT-1)
Brief Title: Efficacy and Safety of Gemcabene in Patients With Homozygous Familial Hypercholesterolemia on Stable, Lipid-Lowering Therapy (COBALT-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-201
Record Dates: First submitted 2016-03-12; First posted 2016-03-30 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Hypercholesteremia
Keywords: LDL-C; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcabene (Experimental): Participants with homozygous familial hypercholesterolemia (HoFH) on stable lipid lowering therapy received 300 milligram (mg) of Gemcabene, orally once daily from day 1 to 28 followed by 600 mg of Gemcabene, orally once daily from day 29 to 56 followed by 900 mg of Gemcabene, orally once daily from day 57 to 84. Participants were followed until Day 112.
  Interventions: Drug: Gemcabene

INTERVENTIONS:
Drug: Gemcabene — 300 mg tablet orally once daily for four weeks followed by 600 mg tablet orally once daily for four weeks followed by 900 mg tablet orally once daily for four weeks.

SUMMARY:
The purpose of this study was to assess the efficacy, safety, and tolerability of multiple doses of Gemcabene in patients with HoFH on stable, lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written and signed informed consent (by patient or legal guardian) prior to any study-specific procedure;
* Male or female ≥17 years of age at time of consent;
* Diagnosis of HoFH by genetic confirmation (including compound heterozygosity) or a clinical diagnosis based on either (1) a history of an untreated LDL-C concentration >500 mg/dL (12.92 mmol/L) together with either appearance of xanthoma before 10 years of age, or evidence of heterozygous familial hypercholesterolemia in both parents or, if history is unavailable, (2) LDL-C >300 mg/dL (7.76 mmol/L) on maximally tolerated lipid-lowering drug therapy;
* Currently on a stable, low-fat, low-cholesterol diet in combination with a pre-existing, regulatory-approved, not excluded lipid-lowering therapy (i.e., statins, monoclonal antibodies to PCSK9, cholesterol absorption inhibitors, bile acid sequestrants, or nicotinic acid, or any combination thereof) at a stable dose for at least 4 weeks prior to the Screening Visit;
* Fasting LDL-C value >130 mg/dL (3.36 mmol/L) at the Screening Visit;
* Physical examination, including vital signs, that is within normal limits or clinically acceptable to the Investigator;
* Weight ≥50 kg;
* Female patients must not be pregnant or lactating. Women of child-bearing potential must have a negative serum pregnancy test at the Screening Visit and negative urine dipstick on Day 1 prior to dosing in order to qualify for the study. Women who are surgically sterile or are clinically confirmed to be post-menopausal (i.e., documented amenorrhea for ≥1 year in the absence of other biological or physiological causes) are not considered to be of child-bearing potential; and
* Women of child-bearing potential must agree to use acceptable methods of contraception throughout the duration of the study and for 30 days after the last dose of study drug. For this study, double-barrier contraception is required.

Exclusion Criteria:

* Other forms of primary hyperlipoproteinemia and secondary causes of hypercholesterolemia (e.g., nephrotic syndrome or hypothyroidism);
* Abnormal liver function test at the Screening Visit (aspartate aminotransferase or alanine aminotransferase >2 × the upper limit of normal [ULN]; total bilirubin >1.5 × ULN; or alkaline phosphatase >2 × ULN based on appropriate age and gender normal values). Patients with bilirubin >1.5 × ULN and history of Gilbert's syndrome may be included; reflexive direct bilirubin testing will be used to confirm Gilbert's syndrome;
* Moderate (Grade B) or severe (Grade C) chronic hepatic impairment according to the Child Pugh classification;
* Active liver disease (e.g., cirrhosis, alcoholic liver disease, hepatitis B virus [HBV], hepatitis C virus [HCV], autoimmune hepatitis, liver failure, liver cancer), history of liver transplant, or known diagnosis of human immunodeficiency virus (HIV);
* Triglycerides value >400 mg/dL (4.52 mmol/L) at the Screening Visit;
* Moderate to severe renal insufficiency defined as an estimated GFR <30 mL/min/1.73m2 (calculated using The Chronic Kidney Disease Epidemiology Collaboration equation) at the Screening Visit;
* Abnormal urinalysis (proteinuria greater than trace or any male or non-menstruating female with greater than trace hematuria), confirmed by reflexive urine protein:creatinine ratio testing;
* Uncontrolled thyroid disease: hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) below the lower limit of normal or >1.5 × ULN, respectively, at the Screening Visit. If controlled, treatment should be stable for at least 3 months prior to the Screening Visit;
* Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (hemoglobin A1c [HbA1c] value >8%), or any diabetic patient taking insulin and/or thiazolidinediones;
* New York Heart Association Class III or IV heart failure;
* Myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, or other major cardiovascular events resulting in hospitalization within 3 months of the Screening Visit. Patients with adequately treated stable angina, per Investigator assessment, may be included;
* Uncontrolled cardiac arrhythmia or prolonged QT on the Screening Visit or Day 1 prior to dosing ECG (QTcF >450 msec for men and >470 msec for women) or known family history of prolonged QT or unexplained sudden cardiac death;
* Uncontrolled hypertension, defined as sitting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg, and confirmed by repeat measurement;
* Currently receiving cancer treatments or, in the Investigator's opinion, at risk of relapse for recent cancer;
* Use of fibrate lipid-lowering agent 6 weeks prior to the Screening Visit;
* Hypersensitivity to or a history of significant adverse reactions to any fibrate lipid lowering agent;
* Use of apheresis (LDL or plasma) 8 weeks prior to the Screening Visit;
* Use of lomitapide 2 months prior to the Screening Visit;
* Use of mipomersen 5 months prior to the Screening Visit;
* Use of any excluded medications or supplements (e.g., potent cytochrome P450 [CYP] 3A4 inhibitors);
* History of drug or alcohol abuse within the past year or inability to comply with protocol requirements, including subject restrictions;
* Previously treated with gemcabene;
* Participation in another clinical study of an investigational agent or device concurrently or within 1 month prior to the Screening Visit, or use of an investigational agent within 1 month or 5 half-lives (if known), whichever is longer, prior to the Screening Visit; or
* Any other finding which, in the opinion of the Investigator, would compromise the patient's safety or participation in the study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Westside Medical Associates of Los Angeles, Beverly Hills, California, United States
- Canada (3):
  - Robarts Research Institute, London, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
- Israel (3):
  - Wolfson Medical Center Internal Medicine Dept., Holon
  - Center for Research, Prevention and Treatment of Atherosclerosis - Cardiology Department of Medicine Kiryat Hadassah, Jerusalem
  - Ziv Medical Center Internal Medicine Department, Safed

REFERENCES:
- [Derived] Gaudet D, Durst R, Lepor N, Bakker-Arkema R, Bisgaier C, Masson L, Golden L, Kastelein JJ, Hegele RA, Stein E. Usefulness of Gemcabene in Homozygous Familial Hypercholesterolemia (from COBALT-1). Am J Cardiol. 2019 Dec 15;124(12):1876-1880. doi: 10.1016/j.amjcard.2019.09.010. Epub 2019 Sep 26. PMID 31685212

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcabene
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All enrolled participants who received at least 1 dose of study drug and had a valid post-baseline efficacy assessment, for a given dose level.
Groups:
- Gemcabene: Participants with homozygous familial hypercholesterolemia (HoFH) on stable lipid lowering therapy received 300 mg of Gemcabene, orally once daily from day 1 to 28 followed by 600 mg of Gemcabene, orally once daily from day 29 to 56 followed by 900 mg of Gemcabene, orally once daily from day 57 to 84.
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: Milligram per deciliter (mg/dL)] — Baseline value was obtained from Friedewald calculation.
  Milligram per deciliter (mg/dL) | 351.25 (181.849)
Non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 379.94 (177.258)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 425.38 (167.058)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 143.56 (62.672)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 45.44 (18.661)
Very low-density lipoprotein cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] | 28.69 (12.530)
High-sensitivity C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: mg/dL] | 5.95 (5.627)
Fibrinogen [Mean (Standard Deviation); unit: mg/dL] | 436.9 (89.23)
Lipoprotein(a) [Mean (Standard Deviation); unit: mg/dL] | 113.5 (92.97)
Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 221.3 (97.25)
Apolipoprotein A-I (ApoA-I) [Mean (Standard Deviation); unit: mg/dL] | 127.9 (46.98)
Apolipoprotein A-II (ApoA-II) [Mean (Standard Deviation); unit: mg/dL] | 30.3 (9.75)
Apolipoprotein C-II (ApoC-II) [Mean (Standard Deviation); unit: mg/dL] | 4.1 (1.21)
Apolipoprotein C-III (ApoC-III) [Mean (Standard Deviation); unit: mg/dL] | 10.6 (4.14)
Apolipoprotein E (ApoE) [Mean (Standard Deviation); unit: mg/dL] | 6.68 (1.738)
LDL-C by Receptor Mutation Status [Mean (Standard Deviation); unit: mg/dL] — Receptor mutation status was categorized as Low density lipoprotein receptor (LDLr) status and European Atherosclerosis Society (EAS) clinical diagnosis of HoFH. Population: FAS Population. Here, number analyzed signifies participants with available data .
  mg/dL
    Negative LDLr: number analyzed (Participants) | 3
    Negative LDLr | 551.33 (105.652)
    Defective LDLr: number analyzed (Participants) | 5
    Defective LDLr | 231.20 (65.191)
    Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
    Met EAS Clinical Diagnosis of HoFH | 374.33 (208.717)
    Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
    Not Met EAS Clinical Diagnosis of HoFH | 282.00 (29.698)
Non-HDL-C by Receptor Mutation Status [Mean (Standard Deviation); unit: mg/dL] — Receptor mutation status was categorized as LDLr status and EAS clinical diagnosis of HoFH. Population: FAS Population. Here, number analyzed signifies participants with available data .
  mg/dL
    Negative LDLr: number analyzed (Participants) | 3
    Negative LDLr | 572.83 (105.419)
    Defective LDLr: number analyzed (Participants) | 5
    Defective LDLr | 264.20 (69.127)
    Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
    Met EAS Clinical Diagnosis of HoFH | 399.92 (205.100)
    Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
    Not Met EAS Clinical Diagnosis of HoFH | 320.00 (5.657)
TC by Receptor Mutation Status [Mean (Standard Deviation); unit: mg/dL] — Receptor mutation status was categorized as LDLr status and EAS clinical diagnosis of HoFH. Population: FAS Population. Here, number analyzed signifies participants with available data .
  mg/dL
    Negative LDLr: number analyzed (Participants) | 3
    Negative LDLr | 601.00 (100.714)
    Defective LDLr: number analyzed (Participants) | 5
    Defective LDLr | 320.00 (82.189)
    Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
    Met EAS Clinical Diagnosis of HoFH | 439.75 (195.112)
    Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
    Not Met EAS Clinical Diagnosis of HoFH | 382.25 (7.425)
TG by Receptor Mutation Status [Mean (Standard Deviation); unit: mg/dL] — Receptor mutation status was categorized as LDLr status and EAS clinical diagnosis of HoFH. Population: FAS Population. Here, number analyzed signifies participants with available data .
  mg/dL
    Negative LDLr: number analyzed (Participants) | 3
    Negative LDLr | 107.67 (9.278)
    Defective LDLr: number analyzed (Participants) | 5
    Defective LDLr | 165.10 (72.694)
    Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
    Met EAS Clinical Diagnosis of HoFH | 128.17 (38.577)
    Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
    Not Met EAS Clinical Diagnosis of HoFH | 189.75 (119.855)
HDL-C by Receptor Mutation Status [Mean (Standard Deviation); unit: mg/dL] — Receptor mutation status was categorized as LDLr status and EAS clinical diagnosis of HoFH. Population: FAS Population. Here, number analyzed signifies participants with available data .
  mg/dL
    Negative LDLr: number analyzed (Participants) | 3
    Negative LDLr | 28.17 (4.726)
    Defective LDLr: number analyzed (Participants) | 5
    Defective LDLr | 55.80 (15.502)
    Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
    Met EAS Clinical Diagnosis of HoFH | 39.83 (17.394)
    Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
    Not Met EAS Clinical Diagnosis of HoFH | 62.25 (13.081)
VLDL-C by Receptor Mutation Status [Mean (Standard Deviation); unit: mg/dL] — Receptor mutation status was categorized as LDLr status and EAS clinical diagnosis of HoFH. Population: FAS Population. Here, number analyzed signifies participants with available data .
  mg/dL
    Negative LDLr: number analyzed (Participants) | 3
    Negative LDLr | 21.50 (1.803)
    Defective LDLr: number analyzed (Participants) | 5
    Defective LDLr | 33.00 (14.530)
    Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
    Met EAS Clinical Diagnosis of HoFH | 25.58 (7.612)
    Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
    Not Met EAS Clinical Diagnosis of HoFH | 38.00 (24.042)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Day 28
Time Frame: Baseline, day 28
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change | -25.54 (8.301)
Statistical Analysis 1: Comparison: Gemcabene; Test type: Other; p = 0.0041, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in LDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used

2. Primary Outcome: Percent Change From Baseline in LDL-C at Day 56
Time Frame: Baseline, day 56
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change | -29.94 (8.301)
Statistical Analysis 1: Comparison: Gemcabene; Test type: Other; p = 0.0010, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Percent Change From Baseline in LDL-C at Day 84
Time Frame: Baseline, day 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change | -29.41 (8.301)
Statistical Analysis 1: Comparison: Gemcabene; Test type: Other; p = 0.0012, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Fasting LDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -82.15 (41.520)
  Day 56 | -99.77 (41.520)
  Day 84 | -94.90 (41.520)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0560, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with Change in LDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0219, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0286, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percent Change From Baseline in Fasting Non-HDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -23.87 (8.105)
  Day 56 | -27.33 (8.105)
  Day 84 | -26.59 (8.105)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0058, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Non-HDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0024, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Fasting Non-HDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -86.64 (44.380)
  Day 56 | -102.89 (44.380)
  Day 84 | -98.26 (44.380)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0592, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Non-HDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0266, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0336, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]

7. Secondary Outcome: Percent Change From Baseline in Fasting Total Cholesterol (TC)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -21.53 (7.287)
  Day 56 | -24.85 (7.287)
  Day 84 | -24.79 (7.287)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0057, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in TC as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0017, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0017, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol (TC)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -91.96 (46.421)
  Day 56 | -108.46 (46.421)
  Day 84 | -104.34 (46.421)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0057, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in TC as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0255, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 86; Test type: Other; p = 0.0312, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -11.99 (15.658)
  Day 56 | -8.37 (15.658)
  Day 84 | -6.55 (15.658)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.4489, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in TG as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 84; Test type: Other; p = 0.5964, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.6785, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in Fasting Triglycerides (TG)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -27.15 (21.615)
  Day 56 | -21.77 (21.615)
  Day 84 | -22.27 (21.615)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300mg: Day 28; Test type: Other; p = 0.2177, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in TG as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600mg: Day 56; Test type: Other; p = 0.3209, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900mg: Day 84; Test type: Other; p = 0.3101, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Percent Change From Baseline in Fasting HDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -11.54 (3.906)
  Day 56 | -12.95 (3.906)
  Day 84 | -12.54 (3.906)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0057, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in HDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0022, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in Fasting HDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -4.80 (1.306)
  Day 56 | -5.05 (1.306)
  Day 84 | -5.55 (1.306)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300mg: Day 28; Test type: Other; p = 0.0008, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in HDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600mg: Day 56; Test type: Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900mg: Day 84; Test type: Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]

13. Secondary Outcome: Percent Change From Baseline in Fasting VLDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -12.84 (15.407)
  Day 56 | -7.79 (15.407)
  Day 84 | -6.55 (15.407)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.4103, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in VLDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.6164, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.6732, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]

14. Secondary Outcome: Change From Baseline in Fasting VLDL-C
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -5.57 (4.261)
  Day 56 | -4.19 (4.261)
  Day 84 | -4.44 (4.261)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300mg: Day 28; Test type: Other; p = 0.2003, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in VLDL-C as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600mg: Day 56; Test type: Other; p = 0.3323, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900mg: Day 84; Test type: Other; p = 0.3047, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]

15. Secondary Outcome: Percent Change From Baseline in Fasting LDL-C as Per Receptor Mutation Status
Description: Receptor mutation status was categorized as LDLr status and EAS clinical diagnosis of HoFH which was reported in this outcome measure.
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -9.78 (10.196)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -14.27 (10.196)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -11.36 (10.196)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -33.97 (6.164)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -38.33 (6.164)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -39.22 (6.164)
  Day 28: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 28: Met EAS Clinical Diagnosis of HoFH | -20.11 (9.502)
  Day 56: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 56: Met EAS Clinical Diagnosis of HoFH | -24.57 (9.502)
  Day 84: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 84: Met EAS Clinical Diagnosis of HoFH | -22.92 (9.502)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -44.40 (4.244)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -48.65 (4.244)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -51.48 (4.244)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.3601, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.1920, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.2912, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0444, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0159, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0235, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

16. Secondary Outcome: Change From Baseline in Fasting LDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -64.16 (67.549)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -92.83 (67.549)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -76.16 (67.549)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -74.43 (40.665)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -85.43 (40.655)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -87.63 (40.655)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -106.54 (312.492)
  Day 56: Met EAS Clinical Diagnosis of HoFH | -125.38 (312.492)
  Day 84: Met EAS Clinical Diagnosis of HoFH | -116.21 (312.492)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -119.38 (15.061)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -133.38 (15.061)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -141.38 (15.061)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.3646, Mixed Models Analysis — Mixed-effects model for repeated measures analysis: Change in LDL-C as dependent variable, visit as fixed effect, patient as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.1994, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.2858, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.0829, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.0492, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.0442, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.7360, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.6917, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.7131, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0009, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]

17. Secondary Outcome: Percent Change From Baseline in Fasting Non-HDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -9.47 (10.497)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -14.21 (10.497)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -11.75 (10.497)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -31.14 (9.861)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -33.83 (9.861)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -34.12 (9.861)
  Day 28: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 28: Met EAS Clinical Diagnosis of HoFH | -18.37 (8.887)
  Day 56: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 56: Met EAS Clinical Diagnosis of HoFH | -21.14 (8.887)
  Day 84: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 84: Met EAS Clinical Diagnosis of HoFH | -19.32 (8.887)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -41.29 (3.577)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -46.81 (3.577)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -49.32 (3.577)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.3880, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.2057, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.2892, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.0052, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.0028, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.0026, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0493, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0253, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0394, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

18. Secondary Outcome: Change From Baseline in Fasting Non-HDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -66.01 (72.386)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -95.34 (72.386)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -80.34 (72.386)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -82.10 (50.684)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -90.50 (50.684)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -92.10 (50.684)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -61.42 (33.020)
  Day 56: Met EAS Clinical Diagnosis of HoFH | -77.08 (33.020)
  Day 84: Met EAS Clinical Diagnosis of HoFH | -68.25 (33.020)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -134.18 (11.456)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -152.18 (11.456)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -160.18 (11.456)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.3833, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.2172, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.2930, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.1217, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.0901, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.0850, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0747, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0279, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0492, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]

19. Secondary Outcome: Percent Change From Baseline in Fasting VLDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28: Met the Genetic Criteria of LDLr: number analyzed (Participants) | 3
  Day 28: Met the Genetic Criteria of LDLr | -2.29 (17.315)
  Day 56: Met the Genetic Criteria of LDLr: number analyzed (Participants) | 3
  Day 56: Met the Genetic Criteria of LDLr | -4.81 (17.315)
  Day 84: Met the Genetic Criteria of LDLr: number analyzed (Participants) | 3
  Day 84: Met the Genetic Criteria of LDLr | -12.19 (17.315)
  Day 28: Not Met the Genetic Criteria of LDLr: number analyzed (Participants) | 5
  Day 28: Not Met the Genetic Criteria of LDLr | -18.82 (30.652)
  Day 56: Not Met the Genetic Criteria of LDLr: number analyzed (Participants) | 5
  Day 56: Not Met the Genetic Criteria of LDLr | -9.22 (30.652)
  Day 84: Not Met the Genetic Criteria of LDLr: number analyzed (Participants) | 5
  Day 84: Not Met the Genetic Criteria of LDLr | -2.82 (30.652)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -8.09 (14.502)
  Day 56: Met EAS Clinical Diagnosis of HoFH | 2.06 (14.502)
  Day 84: Met EAS Clinical Diagnosis of HoFH | 2.72 (14.502)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -15.53 (3.488)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -25.75 (3.488)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -22.80 (3.488)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.8972, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.7867, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.4974, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.5464, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.7668, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.9276, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.5821, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.8881, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.8525, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0112, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0028, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]

20. Secondary Outcome: Change From Baseline in Fasting VLDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28: Met the Genetic Criteria of LDLr: number analyzed (Participants) | 3
  Day 28: Met the Genetic Criteria of LDLr | -0.50 (3.821)
  Day 56: Met the Genetic Criteria of LDLr: number analyzed (Participants) | 3
  Day 56: Met the Genetic Criteria of LDLr | -1.17 (3.821)
  Day 84: Met the Genetic Criteria of LDLr: number analyzed (Participants) | 3
  Day 84: Met the Genetic Criteria of LDLr | -2.83 (3.821)
  Day 28: Not Met the Genetic Criteria of LDLr: number analyzed (Participants) | 5
  Day 28: Not Met the Genetic Criteria of LDLr | -8.55 (6.869)
  Day 56: Not Met the Genetic Criteria of LDLr: number analyzed (Participants) | 5
  Day 56: Not Met the Genetic Criteria of LDLr | -5.95 (6.869)
  Day 84: Not Met the Genetic Criteria of LDLr: number analyzed (Participants) | 5
  Day 84: Not Met the Genetic Criteria of LDLr | -5.35 (6.869)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -2.18 (29.378)
  Day 56: Met EAS Clinical Diagnosis of HoFH | 0.98 (29.378)
  Day 84: Met EAS Clinical Diagnosis of HoFH | 0.65 (29.378)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -1.55 (1.816)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -5.55 (1.816)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -5.55 (1.816)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.8985, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.7664, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.4755, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.2286, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.3975, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.4460, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9414, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9735, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9825, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.4420, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0378, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0378, Mixed Models Analysis — [p-value comment as in outcome 14, analysis 1]

21. Secondary Outcome: Percent Change From Baseline in Fasting HDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -18.44 (14.443)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -20.63 (14.443)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -6.75 (14.443)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -9.51 (3.507)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -10.45 (3.507)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -18.12 (3.507)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -11.92 (5.805)
  Day 56: Met EAS Clinical Diagnosis of HoFH | -15.77 (5.805)
  Day 84: Met EAS Clinical Diagnosis of HoFH | -15.69 (5.805)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -16.98 (3.417)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -11.07 (3.417)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -9.67 (3.417)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.2305, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.1836, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.6501, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.0139, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.0077, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0507, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0118, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0122, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0077, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0317, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0473, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]

22. Secondary Outcome: Change From Baseline in Fasting HDL-C as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28: NegativeLDLr: number analyzed (Participants) | 3
  Day 28: NegativeLDLr | -4.96 (3.738)
  Day 56: NegativeLDLr: number analyzed (Participants) | 3
  Day 56: NegativeLDLr | -5.29 (3.738)
  Day 84: NegativeLDLr: number analyzed (Participants) | 3
  Day 84: NegativeLDLr | -1.62 (3.738)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -5.19 (1.508)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -5.39 (1.508)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -8.39 (1.508)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -4.16 (1.755)
  Day 56: Met EAS Clinical Diagnosis of HoFH | -5.50 (1.755)
  Day 84: Met EAS Clinical Diagnosis of HoFH | -6.50 (1.755)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -9.07 (1.867)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -6.07 (1.867)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -5.07 (1.867)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.2143, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.1874, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.6731, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.0027, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.0020, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0258, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0044, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0083, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0314, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0533, Mixed Models Analysis — [p-value comment as in outcome 12, analysis 1]

23. Secondary Outcome: Percent Change From Baseline in Fasting TC as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -10.02 (10.577)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -14.57 (10.577)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -11.64 (10.577)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -26.43 (9.116)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -29.01 (9.116)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -30.67 (9.116)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -17.30 (8.845)
  Day 56: Met EAS Clinical Diagnosis of HoFH | -20.39 (8.845)
  Day 84: Met EAS Clinical Diagnosis of HoFH | -19.69 (8.845)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -38.47 (2.496)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -42.48 (2.496)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -44.31 (2.496)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.3657, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.1983, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.2970, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.0092, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.0049, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.0033, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0618, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0298, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0352, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]

24. Secondary Outcome: Change From Baseline in Fasting TC as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -70.92 (75.095)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -100.58 (75.095)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -81.92 (75.095)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -84.61 (57.378)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -93.21 (57.378)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -97.81 (57.378)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -65.58 (33.715)
  Day 56: Met EAS Clinical Diagnosis of HoFH | -82.58 (33.715)
  Day 84: Met EAS Clinical Diagnosis of HoFH | -74.75 (33.715)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -143.67 (9.885)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -158.67 (9.885)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -165.67 (9.885)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr; Test type: Other; p = 0.3672, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.2101, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.3009, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.1567, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.1207, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.1045, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0631, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0217, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0359, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]

25. Secondary Outcome: Percent Change From Baseline in Fasting TG as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -1.30 (17.390)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -5.17 (17.390)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -11.36 (17.390)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -17.89 (32.682)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -9.77 (32.682)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -3.14 (32.682)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -7.02 (14.510)
  Day 56: Met EAS Clinical Diagnosis of HoFH | 1.43 (14.510)
  Day 84: Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 6
  Day 84: Met EAS Clinical Diagnosis of HoFH | 2.98 (14.510)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -15.72 (3.302)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -26.60 (3.302)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -23.96 (3.302)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.9417, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.7722, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.5283, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.5905, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.7682, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.9245, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.6325, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9221, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.8387, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0089, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0013, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]

26. Secondary Outcome: Change From Baseline in Fasting TG as Per Receptor Mutation Status
Description: as for outcome 15
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, number analyzed signifies those participants who were evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28: Negative LDLr: number analyzed (Participants) | 3
  Day 28: Negative LDLr | -2.00 (19.308)
  Day 56: Negative LDLr: number analyzed (Participants) | 3
  Day 56: Negative LDLr | -6.33 (19.308)
  Day 84: Negative LDLr: number analyzed (Participants) | 3
  Day 84: Negative LDLr | -13.33 (19.308)
  Day 28: Defective LDLr: number analyzed (Participants) | 5
  Day 28: Defective LDLr | -41.94 (35.093)
  Day 56: Defective LDLr: number analyzed (Participants) | 5
  Day 56: Defective LDLr | -30.74 (35.093)
  Day 84: Defective LDLr: number analyzed (Participants) | 5
  Day 84: Defective LDLr | -27.34 (35.093)
  Day 28: Met EAS Clinical Diagnosis of HoFH | -10.33 (102.229)
  Day 56: Met EAS Clinical Diagnosis of HoFH | 3.83 (102.229)
  Day 84: Met EAS Clinical Diagnosis of HoFH | 3.17 (102.229)
  Day 28: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 28: Not Met EAS Clinical Diagnosis of HoFH | -7.82 (8.738)
  Day 56: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 56: Not Met EAS Clinical Diagnosis of HoFH | -28.82 (8.738)
  Day 84: Not Met EAS Clinical Diagnosis of HoFH: number analyzed (Participants) | 2
  Day 84: Not Met EAS Clinical Diagnosis of HoFH | -28.82 (8.738)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Negative LDLr); Test type: Other; p = 0.9195, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Negative LDLr); Test type: Other; p = 0.7497, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Negative LDLr); Test type: Other; p = 0.5056, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Defective LDLr); Test type: Other; p = 0.2468, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Defective LDLr); Test type: Other; p = 0.3920, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Defective LDLr); Test type: Other; p = 0.4456, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9203, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9704, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.9755, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene; Gemcabene 300 mg: Day 28 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.4213, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 11: Comparison: Gemcabene; Gemcabene 600 mg: Day 56 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0300, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 12: Comparison: Gemcabene; Gemcabene 900 mg: Day 84 (Not Met EAS Clinical Diagnosis of HoFH); Test type: Other; p = 0.0300, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]

27. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥15%
Time Frame: Days 28, 56 and 84
Population: FAS Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Participants
  Day 28 | 6
  Day 56 | 6
  Day 84 | 7

28. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥20%
Time Frame: Days 28, 56 and 84
Population: FAS Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Participants
  Day 28 | 5
  Day 56 | 6
  Day 84 | 6

29. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥25%
Time Frame: Days 28, 56 and 84
Population: FAS Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Participants
  Day 28 | 5
  Day 56 | 5
  Day 84 | 5

30. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥30%
Time Frame: Days 28, 56 and 84
Population: FAS Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Participants
  Day 28 | 4
  Day 56 | 5
  Day 84 | 4

31. Secondary Outcome: Number of Participants Achieving an LDL-C Value <100 mg/dL (2.59 mmol/L)
Time Frame: Days 28, 56 and 84
Population: FAS Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Participants
  Day 28 | 1
  Day 56 | 1
  Day 84 | 1

32. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (hsCRP)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | 63.11 (26.022)
  Day 56 | -26.67 (26.022)
  Day 84 | -16.89 (26.022)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300mg: Day 28; Test type: Other; p = 0.0294, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in hsCRP as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.3228, Mixed Models Analysis — [p-value comment as in outcome 32, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.5268, Mixed Models Analysis — [p-value comment as in outcome 32, analysis 1]

33. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/L
  Day 28 | 5.30 (3.105)
  Day 56 | -1.91 (3.105)
  Day 84 | 0.46 (3.105)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.1099, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in hsCRP as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.5478, Mixed Models Analysis — [p-value comment as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.8837, Mixed Models Analysis — [p-value comment as in outcome 33, analysis 1]

34. Secondary Outcome: Percent Change From Baseline in Fibrinogen
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | 8.20 (3.985)
  Day 56 | -6.08 (3.985)
  Day 84 | -5.09 (3.985)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0587, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in fibrinogen as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.1491, Mixed Models Analysis — [p-value comment as in outcome 34, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.2224, Mixed Models Analysis — [p-value comment as in outcome 34, analysis 1]

35. Secondary Outcome: Change From Baseline in Fibrinogen
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | 34.17 (19.141)
  Day 56 | -34.58 (19.141)
  Day 84 | -28.46 (19.141)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0959, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in fibrinogen as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0923, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.1592, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]

36. Secondary Outcome: Percent Change From Baseline in Fasting Lipoprotein(a)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | 6.90 (12.362)
  Day 56 | 5.84 (12.362)
  Day 84 | 15.62 (12.362)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.5856, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Lipoprotein(a) as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.6440, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.2269, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]

37. Secondary Outcome: Change From Baseline in Fasting Lipoprotein(a)
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
nmol/L
  Day 28 | 19.39 (26.804)
  Day 56 | 18.51 (26.804)
  Day 84 | 21.51 (26.804)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.4814, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Lipoprotein(a) as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.5011, Mixed Models Analysis — [p-value comment as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.4356, Mixed Models Analysis — [p-value comment as in outcome 37, analysis 1]

38. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein B
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -17.95 (9.034)
  Day 56 | -23.98 (9.034)
  Day 84 | -21.58 (9.034)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0669, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Apolipoprotein B as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0189, Mixed Models Analysis — [p-value comment as in outcome 38, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0316, Mixed Models Analysis — [p-value comment as in outcome 38, analysis 1]

39. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein B
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -39.24 (19.882)
  Day 56 | -57.87 (19.882)
  Day 84 | -49.37 (19.882)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0685, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Apolipoprotein B as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0114, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0263, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 1]

40. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-I
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -6.27 (4.082)
  Day 56 | -3.86 (4.082)
  Day 84 | -8.06 (4.082)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.1466, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Apolipoprotein A-I as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.3598, Mixed Models Analysis — [p-value comment as in outcome 40, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0685, Mixed Models Analysis — [p-value comment as in outcome 40, analysis 1]

41. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein A-I
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -7.26 (4.967)
  Day 56 | -4.88 (4.967)
  Day 84 | -11.88 (4.967)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.1660, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Apolipoprotein A-I as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.3423, Mixed Models Analysis — [p-value comment as in outcome 41, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0313, Mixed Models Analysis — [p-value comment as in outcome 41, analysis 1]

42. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-II
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | 2.00 (5.473)
  Day 56 | 4.41 (5.473)
  Day 84 | 1.97 (5.473)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.7196, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Apolipoprotein A-II as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.4343, Mixed Models Analysis — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.7241, Mixed Models Analysis — [p-value comment as in outcome 42, analysis 1]

43. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein A-II
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | 0.38 (1.423)
  Day 56 | 1.00 (1.423)
  Day 84 | 0.25 (1.423)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.7952, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Apolipoprotein A-II as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.4931, Mixed Models Analysis — [p-value comment as in outcome 43, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.8622, Mixed Models Analysis — [p-value comment as in outcome 43, analysis 1]

44. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein C-II
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population. Here, overall number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure only.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 7
Percent Change
  Day 28 | -1.69 (74.431)
  Day 56 | 8.31 (74.431)
  Day 84 | 21.64 (74.431)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.9823, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Apolipoprotein C-II as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.9129, Mixed Models Analysis — [p-value comment as in outcome 44, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 600 mg: Day 84; Test type: Other; p = 0.7762, Mixed Models Analysis — [p-value comment as in outcome 44, analysis 1]

45. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein C-II
Time Frame: Baseline, days 28, 56 and 84
Population: as for outcome 44
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 7
mg/dL
  Day 28 | 0.71 (0.615)
  Day 56 | 1.14 (0.615)
  Day 84 | 1.71 (0.615)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.2683, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Apolipoprotein C-II as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0880, Mixed Models Analysis — [p-value comment as in outcome 45, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0165, Mixed Models Analysis — [p-value comment as in outcome 45, analysis 1]

46. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein C-III
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -8.86 (11.616)
  Day 56 | -10.71 (11.616)
  Day 84 | -7.47 (11.616)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.4585, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Apolipoprotein C-III as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.3721, Mixed Models Analysis — [p-value comment as in outcome 46, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.5305, Mixed Models Analysis — [p-value comment as in outcome 46, analysis 1]

47. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein C-III
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -1.37 (1.260)
  Day 56 | -1.62 (1.260)
  Day 84 | -1.37 (1.260)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.2937, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Apolipoprotein C-III as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.2182, Mixed Models Analysis — [p-value comment as in outcome 47, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.2937, Mixed Models Analysis — [p-value comment as in outcome 47, analysis 1]

48. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein E
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
Percent Change
  Day 28 | -19.57 (8.699)
  Day 56 | -23.01 (8.699)
  Day 84 | -19.20 (8.699)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0411, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with percent change in Apolipoprotein E as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0192, Mixed Models Analysis — [p-value comment as in outcome 48, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0445, Mixed Models Analysis — [p-value comment as in outcome 48, analysis 1]

49. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein E
Time Frame: Baseline, days 28, 56 and 84
Population: FAS Population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 8
mg/dL
  Day 28 | -1.40 (0.641)
  Day 56 | -1.65 (0.641)
  Day 84 | -1.45 (0.641)
Statistical Analysis 1: Comparison: Gemcabene; Gemcabene 300 mg: Day 28; Test type: Other; p = 0.0465, Mixed Models Analysis — Mixed-effects model for repeated measures analysis with change in Apolipoprotein E as dependent variable, visit as fixed effect, participant as a random effect. Auto-regressive variance-covariance structure was used
Statistical Analysis 2: Comparison: Gemcabene; Gemcabene 600 mg: Day 56; Test type: Other; p = 0.0221, Mixed Models Analysis — [p-value comment as in outcome 49, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene; Gemcabene 900 mg: Day 84; Test type: Other; p = 0.0402, Mixed Models Analysis — [p-value comment as in outcome 49, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Up to 112 days)
Groups:
- Gemcabene 300 mg: Participants with homozygous familial hypercholesterolemia (HoFH) on stable lipid lowering therapy received 300 mg of Gemcabene, orally once daily from day 1 to 28.
- Gemcabene 600 mg: Participants with homozygous familial hypercholesterolemia (HoFH) on stable lipid lowering therapy received 600 mg of Gemcabene, orally once daily from day 29 to 56.
- Gemcabene 900 mg: Participants with homozygous familial hypercholesterolemia (HoFH) on stable lipid lowering therapy received 900 mg of Gemcabene, orally once daily from day 57 to 84.
Arm/Group | Gemcabene 300 mg | Gemcabene 600 mg | Gemcabene 900 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 4/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcabene 300 mg (N=8) | Gemcabene 600 mg (N=8) | Gemcabene 900 mg (N=8)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Energy increased (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0
Myoglobinuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT02722408/SAP_000.pdf
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT02722408/Prot_001.pdf